CLINICAL TRIAL: NCT07319754
Title: The Effect of Transcutaneous Electrical Nerve Stimulation (TENS) on Postoperative Pain and Sleep After Inguinal Hernia Surgery: A Randomized Controlled Trial
Brief Title: TENS for Pain and Sleep After Hernia Surgery
Acronym: TENS-HERNIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Abdurrahman Acar, Research Assistant, Faculty of Health Sciences, Niğde Ömer Halisdemir University, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22504254-050.04-NOHU; SAT 2025/15-BAGEP (Other: Niğde Ömer Halisdemir University Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2025-12-10; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Inguinal Hernia; Postoperative Pain; Sleep Disturbance
Keywords: Inguinal hernia; Postoperative Pain; Sleep Disturbance; Transcutaneous Electrical Nerve Stimulation (TENS)
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Parasomnias | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups. The intervention group will receive physician-supervised Transcutaneous Electrical Nerve Stimulation (TENS) following inguinal hernia surgery, while the control group will receive standard postoperative care without TENS. Outcomes will be compared between groups to evaluate the effect of TENS on postoperative pain and sleep quality.
Masking Description: No additional parties are masked in this study. The trial is conducted as open label, and both participants and investigators are aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): TENS Group (Experimental): Participants in this arm will receive physician-supervised Transcutaneous Electrical Nerve Stimulation (TENS) following inguinal hernia surgery. TENS will be applied to the inguinal region using surface electrodes according to a standardized protocol. The intervention aims to reduce postoperative pain and improve sleep quality compared with standard care.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Arm 2: Standard Care Group (Active Comparator): Participants in this arm will receive standard postoperative care following inguinal hernia surgery, without TENS application. Outcomes will be assessed in the same way as the experimental group for comparison.
  Interventions: Other: Standard Postoperative Care

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Physician-supervised application of TENS to the inguinal region after hernia surgery, following a standardized protocol.
  Arms: Arm 1 (Experimental): TENS Group
Other: Standard Postoperative Care — Participants in this arm will receive routine postoperative care following inguinal hernia surgery, without TENS application.
  Arms: Arm 2: Standard Care Group

SUMMARY:
This study evaluates whether Transcutaneous Electrical Nerve Stimulation (TENS) improves postoperative pain and sleep quality in adults undergoing inguinal hernia surgery. After surgery, participants will receive physician-supervised TENS or usual care. Pain intensity and sleep quality will be measured and compared between groups to assess the effectiveness and safety of TENS as a supportive recovery method.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the effects of Transcutaneous Electrical Nerve Stimulation (TENS) on postoperative pain and sleep quality in patients undergoing inguinal hernia repair. Inguinal hernia is one of the most common surgical conditions worldwide, with increasing prevalence in recent years. Although tension-free herniorrhaphy has become the gold standard technique due to its low recurrence rate, rapid recovery, and cost-effectiveness, chronic postoperative inguinal pain (CPIP) remains a significant complication that negatively affects quality of life. CPIP is typically defined as new or altered groin pain persisting for more than three months after surgery, and its pathophysiology is not fully understood. Nerve injury or entrapment of the ilioinguinal, iliohypogastric, or genitofemoral nerves is considered a major contributor.

Postoperative pain management often relies on opioid analgesics, which carry risks of dependence, respiratory depression, and prolonged hospitalization. Therefore, non-pharmacological alternatives are of growing interest. TENS is a minimally invasive neuromodulation technique that modulates pain signals, most commonly explained by the Gate Control Theory, in which stimulation of large myelinated fibers inhibits transmission of pain through smaller nociceptive fibers. Previous studies have suggested potential benefits of TENS in CPIP, but evidence remains limited and inconsistent. Moreover, chronic pain is frequently associated with sleep disturbances, further impairing physical and psychological well-being. TENS may therefore improve both pain and sleep quality in this patient population.

The study will be conducted between October 2025 and October 2026 at the General Surgery Department of SBÜ Adana City Training and Research Hospital. Eligible participants will be adults (≥18 years) undergoing inguinal hernia surgery who are conscious, cooperative, and without contraindications to TENS. Exclusion criteria include cardiac pacemakers or implanted electronic devices, uncontrolled epilepsy or neurological disorders, chronic opioid use prior to surgery, severe psychiatric or cognitive impairment, dermatological conditions at electrode sites, requirement for additional analgesic/regional block during follow-up, or concurrent participation in another clinical trial.

Sample size was determined by power analysis, requiring 40 patients in the intervention group and 40 in the control group (total n=80) to detect a significant difference with α=0.05 and power=0.80. Data collection will include a Personal Information Form, the Visual Analog Scale (VAS) for pain intensity, and the Richards-Campbell Sleep Questionnaire (RCSQ) for sleep quality. VAS is a validated, simple, and widely used tool for assessing subjective pain intensity, while the RCSQ evaluates multiple dimensions of sleep quality using visual analog scales.

The primary hypothesis is that TENS will reduce postoperative pain and improve sleep quality compared with standard care. The null hypothesis states that TENS has no effect on these outcomes. Ethical approval has been obtained, and all procedures will be performed under physician supervision to ensure patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) undergoing elective inguinal hernia surgery

Ability to provide informed consent

Willingness to comply with study procedures

Exclusion Criteria:

* History of epilepsy, cardiac pacemaker, or other contraindications to TENS

Severe psychiatric or neurological disorders affecting pain or sleep assessment

Allergy or intolerance to electrode materials

Patients requiring emergency surgery

Inability to complete questionnaires (VAS, PSQI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | First 24 hours after surgery
  Pain intensity will be measured using the Visual Analog Scale (VAS) at 6, 12, and 24 hours postoperatively.
Change in Pain Intensity (VAS) | First 24 hours after surgery
  Pain intensity will be measured using the Visual Analog Scale (VAS) at 6, 12, and 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.